CLINICAL TRIAL: NCT01240330
Title: Evaluation of the Effect of the Vasculaire Compression System on Flow Velocity in the Femoral Vein
Brief Title: Vasculaire Compression System Increases Flow Velocity in the Femoral Vein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venous Health Systems, Inc. (Industry)
Responsible Party: Thomas J. Fogarty, M.D. Principal Investigator, Venous Health Systems, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VenousHealth-001
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Venous Thrombosis
Keywords: Deep Vein Thrombosis; Effects of compression therapy; Peak Flow Velocity
MeSH Terms: conditions — Venous Thrombosis | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pneumatic Compression therapy — Subject comparison analysis of femoral venous Peak Flow Velocity at rest and during compression therapy.
  Other Names: Intermittent pneumatic compression; Sequential compression

SUMMARY:
The objective of this clinical study was to demonstrate the performance of the Vasculaire Compression System to increase femoral venous peak velocity (PFV) in healthy subjects. This study was a single-arm, open label, prospective, single-center clinical study.

DETAILED DESCRIPTION:
Venous thromboembolism, e.g. deep vein thrombosis (DVT) and pulmonary embolism, occurs in approximately one in 1,000 persons in the United States annually and results in more than 250,000 hospital admissions annually in the United States. Intermittent pneumatic compression (IPC), which prevents stasis in the lower limbs, has been shown to be a safe and effective method of prophylaxis of DVT in studies comparing the incidence of DVT and pulmonary embolism with and without IPC. IPC devices decrease venous stasis by augmenting the venous blood flow in the lower extremities. Studies have suggested that an important indicator of the effectiveness of an IPC device in preventing DVT is the peak femoral venous velocity augmentation during the compression phase as compared with the decompression phase of the device.

IPC devices produced in the early 1980s and 1990s were cumbersome, noisy and required external power sources, making them suitable only for non-ambulatory patients. Furthermore, these devices have been associated with poor compliance in trauma patients in a hospital setting, and the poor compliance was associated with a higher rate of DVT.

The aim of this study is to test the hemodynamic performance of a new portable IPC device, the Venous Health Systems' Vasculaire Compression System. This new device is designed to provide patient comfort and convenience of use while providing similar improvement in venous blood flow when compared with existing IPC devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 years old and 65 years old;
* Capable of and willing to lay supine for approximately one hour;
* Subjects must provide written informed consent

Exclusion Criteria:

* History of Deep Vein Thrombosis (DVT) or suspected DVT;
* History of vascular disease, e.g. coronary or peripheral artery disease;
* History of stroke;
* History of pulmonary edema;
* History of congestive heart failure;
* Diabetes mellitus;
* Past or present smoker;
* Surgery or trauma to the right leg within the last six months;
* Open ulcers or wounds on the right leg;
* Pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Fogarty, M.D., Principal Investigator — Founder
Locations (1):
- Venous Health System, Inc., Portola Valley, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Duration: 4 days First subject enrolled: August 31, 2010 Last subject completed: September 3, 2010
Pre-assignment Details: No enrolled participants were excluded from the study.
Groups:
- Pneumatic Compression Therapy: The Vasculaire System provided compression therapy to the foot and calf of the participant's right leg. The system compressed and released the foot and calf to increase blood flow and circulation of the participant's right limb. Ten cycles of compression therapy was applied. Increase in blood flow rate was measured in the participants femoral vein using duplex ultrasonography.
Period: Overall Study
Arm/Group | Pneumatic Compression Therapy
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pneumatic Compression Therapy
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 (0)
  Between 18 and 65 years | 33 (5.20)
  >=65 years | 0 (0)
Age Continuous [Mean (Standard Deviation); unit: years] | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Femoral Venous Peak Flow Velocity Compared to Resting Baseline
Description: The femoral vein in the mid-thigh area was located and the femoral venous Peak Flow Velocity (PFV)was measured using duplex ultrasound during the compression phase of treatment. PFV is the maximum velocity of blood flow achieved when the foot and calf compression is applied. The PFV was then compared to the subject's own baseline PFV using a paired t-test.
Time Frame: 3 measurements/10 min. therapy
Measure: Mean (95% Confidence Interval); unit: cm/s
Arm/Group | Pneumatic Compression Therapy
Number analyzed (Participants) | 33
cm/s | 18.9 [16.3 to 21.6]
Statistical Analysis 1: Comparison: Pneumatic Compression Therapy; The femoral venous peak flow velocity (PFV) compared to the subject's own resting baseline PFV; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean Difference (Final Values) = 18.9, 95% CI 2-sided [16.30 to 21.59], Standard Deviation 7.46

2. Secondary Outcome: PFV Percent Augmentation
Description: Peak Flow Velocity (PFV) from the compression phase subtracted from the PFV from the decompression phase divided by the PFV from the decompression phase expressed as the percent augmentation.
Time Frame: 3 measurements/10 minute therapy
Measure: Mean (Standard Deviation); unit: percentages
Arm/Group | Pneumatic Compression Therapy
Number analyzed (Participants) | 33
percentages
  PFV Percent Augmentation | 175.5 (71.7)

3. Secondary Outcome: Subject Comfort
Description: Subject comfort was measured on a scale 1 to 5 (1=negative response; 5=positive response) during the sleeve installation, during use, and completion.
Time Frame: 10 min therapy
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Pneumatic Compression Therapy
Number analyzed (Participants) | 33
Units on a Scale
  Comfort during installation | 4.94 (0.24)
  Comfort during use | 4.94 (0.24)
  Comfort after completion | 5.00 (0)

ADVERSE EVENTS:
Arm/Group | Pneumatic Compression Therapy
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No